CLINICAL TRIAL: NCT00244166
Title: Threecenter Placebo Controlled Three Arm Trial in Patients With Active Ankylosing Spondylitis With Prednisolone
Brief Title: Prednisolone in Active Ankylosing Spondylitis (AS)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-01
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Ankylosing Spondylitis
Keywords: treatment; ankylosing spondylitis; prednisolone; trial; steroid
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Prednisolone

INTERVENTIONS:
Drug: prednisolone

SUMMARY:
1. to investigate whether steroids are effective in ankylosing spondylitis
2. if steroids are effective to describe how quick they work

DETAILED DESCRIPTION:
Treatment of inflammatory rheumatic conditions with glucocorticosteroids is a mainstay in therapy. In rheumatic diseases such as rheumatoid arthritis, systemic lupus erythematodes and polymyalgia rheumatica glucocorticosteroids show a prompt effect in regards of musculoskeletal symptoms.

Ankylosing spondylitis (AS) is an inflammatory rheumatic disease mainly affecting the spine. However peripheral joints, entheses and the eyes can also be affected. The rheumatic symptoms of AS patients typically show good and quick response to treatment with nonsteroidal antirheumatic drugs (NSAIDs). In contrast to rheumatoid arthritis there is no proof that disease modifying antirheumatic drugs (DMARDs) work. Surprisingly there is the common opinion, mainly based on personal experiences, that glucocorticosteroids in spondylarthropathies do not work. However there are no reliable clinical studies answering this question. In the literature of the last 20 years there are only single reports about the treatment of AS with highly dosed methylprednisolone (intravenous pulse therapy). The pretended lack of effectiveness of glucocorticosteroids surprises moreover as NSAIDs are very effective as well as local intraarticular steroid injections including the sacroiliac joints. In addition with magnetic resonance imaging acute inflammatory lesions can be visualized especially as subchondral edema in bone marrow. Besides about 70% of patients with active AS show elevated inflammatory serum markers such as erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP). Moreover we could recently that a treatment of AS patients with the monoclonal antibody against TNFa (Infliximab) is highly effective. TNFa is a very important pro-inflammatory cytokine (Brandt et al 2000).

For all these reasons it is very important and urgent to perform a study for the treatment of active AS with glucocorticosteroids using evaluated measuring instruments.

ELIGIBILITY:
Inclusion Criteria:

1. ankylosing spondylitis according to the modified NY criteria 1984
2. age between 18 and 70 years
3. insufficient response to therapy with NSAIDs
4. BASDAI > 4
5. Previous therapy with DMARDs (such as sulfasalazine, methotrexate etc.) or steroids less than or equal to 7,5mg is allowed, should be discontinued or stable 4 weeks before study start
6. written informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. current severe infection or during the last 3 months
3. suspected opportunistic infection during the past 2 months (such as Herpes zoster, cytomegaly-, Pneumocystis carinii-infection), HIV-infection
4. Malignancies
5. severe cardial, renal, hematological, endocrinological, pulmonal, gastrointestinal (such as peptic ulcers) neurological, hepatic (viral or toxic hepatitis) concomitant disease, uncontrolled arterial hypertension remitting thrombosis, embolism
6. Diabetes mellitus or increased blood glucose test
7. uncontrolled glaucoma
8. active immunization during the past 2 weeks or planned for the next 8 weeks
9. pathologic laboratory test results: creatinine >200 µmol/l, liver enzymes > 2,5 fold, AP >2,5 fold upper normal ranges
10. significant pathological changes during physical examination
11. clinical trial participation during the past 30 days before screening
12. intake of "hard drugs" (such as cocaine, heroin)
13. therapy with more than 7,5 mg prednisolone, intraarticular steroids during the past 4 weeks before study start
14. current application for retirement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2002-05; Study Completion 2008-08

PRIMARY OUTCOMES:
50% improvement of BASDAI after 14 days of treatment

SECONDARY OUTCOMES:
Improvement of pain on a VAS 0 - 10
Decrease of CRP/ BSG
Number of swollen/tender joints
number of enthesitic localisations
improvement of function (BASFI)
improvement of quality of life (SF12)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, Prof., Principal Investigator — Charité Campus Benjamin-Franklin Rheumatology
Locations (3):
- Germany (3):
  - Charité Campus Benjamin-Franklin Rheumatolgy, Berlin
  - Immanuel Hospital Rheumatology, Berlin
  - Rheumazentrum Ruhrgebiet, Herne

REFERENCES:
- [Derived] Haibel H, Fendler C, Listing J, Callhoff J, Braun J, Sieper J. Efficacy of oral prednisolone in active ankylosing spondylitis: results of a double-blind, randomised, placebo-controlled short-term trial. Ann Rheum Dis. 2014 Jan;73(1):243-6. doi: 10.1136/annrheumdis-2012-203055. Epub 2013 Apr 26. PMID 23625982